CLINICAL TRIAL: NCT04852029
Title: Prospective Assessment of Impact of Personalized Dosing of Low-dose Human Chorionic Gonadotropin (hCG) on in Vitro Fertilization (IVF) Outcomes
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: recruitment issues
Sponsor: Reproductive Medicine Associates of New Jersey (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: RMA-2021-01
Record Dates: First submitted 2021-04-15; First posted 2021-04-21 (Actual); Last update posted 2022-01-28 (Actual); Status verified 2022-01

CONDITIONS: Infertility, Female
MeSH Terms: conditions — Infertility, Female

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control Group (Active Comparator): to remain on current dose of low dose hCG
  Interventions: Other: Low dose hCG
- Intervention Group (Experimental): increased dose of low dose hCG prescribed
  Interventions: Other: Low dose hCG

INTERVENTIONS:
Other: Low dose hCG — Patients will either maintain the current dose of have an increased dose prescribed based on randomization

SUMMARY:
The purpose of the study is to determine the effect of tailoring dosage of low-dose hCG secondary to serum hCG levels during IVF ovarian stimulation on sustained implantation rates of preimplantation genetically tested euploid embryos.

DETAILED DESCRIPTION:
The objective of this study is to conduct a double-blind prospective randomized control trial to determine if individualized hCG titration based on a patient's serum hCG level above or below the predetermined serum hCG level improves IVF outcomes, primarily sustained implantation rates. Patients who fall below the desired serum hCG threshold will be randomized to either maintaining their current dose of low dose hCG or being increased.

ELIGIBILITY:
Inclusion Criteria:

1. Patients whose physicians plan to prescribe low-dose hCG for ovarian stimulation
2. Age 18-46
3. Negative serum hCG prior to start of COH
4. BMI >18 and <35
5. Plan for ejaculated sperm use
6. Plan for PGT testing with euploid embryo transfer

Exclusion Criteria:

1. Administration of low-dose hCG during frozen embryo transfer cycle
2. Concomitant Menopur administration during ovarian stimulation or during frozen embryo transfer cycle
3. BMI <18 or >35
4. Age <18 or >46
5. Presence of hydrosalpinxes that communicate with the endometrial cavity
6. Diagnosis of endometrial insufficiency: prior cycle with maximal endometrial thickness ≤ 6mm, abnormal endometrial pattern (failure to attain a trilaminar appearance), and persistent endometrial fluid
7. Uncorrected uterine factor infertility (uterine anomaly, submucosal myomas, uterine septum)
8. Male partner with <100,000 total motile spermatozoa per ejaculate (donor sperm is acceptable)
9. Use of surgical procedures to obtain sperm
10. Couples undergoing IVF for fertility preservation with no immediate plan for subsequent FET (embryo banking)
11. Personal history of repeated pregnancy loss (two or more unexplained clinical losses defined by presence of fetal heartbeat)
12. Declination of PGT testing

Ages: 18 Years to 46 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2021-08-16 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
sustained implantation rate | 8 weeks gestational age
  presence of fetal heart beat upon discharge

CONTACTS AND LOCATIONS:
Locations (1):
- Reproductive Medicine Associates of New Jersey, Basking Ridge, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No